CLINICAL TRIAL: NCT03589378
Title: Efficacy of PEAF for Septic Shock With Multiple Organ Dysfunction Syndrome in ICU:A Multicenter,Open-Parallelled ,Randomized and Controlled Clinical Trial
Brief Title: Therapeutic Plasma Exchange Adsorption Diafiltration
Acronym: PEAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZLY2017007; 20173357201815 (Other Grant/Funding Number: ShenZhen Second People's Hospital)
Record Dates: First submitted 2018-04-22; First posted 2018-07-17 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Septic Shock; Multiple Organ Dysfunction Syndrome
MeSH Terms: conditions — Shock, Septic; Multiple Organ Failure

STUDY DESIGN:
Intervention Model Description: a Multicenter,Randomized and Controlled Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEAF (Experimental): Intervention group:the patient will receive treatment with PEAF immediately after randomization.PEAF that is TPE (20ml/kg/d Fresh frozen plasma, Blood pump: 120ml/min, replacement pump 20ml/kg/min, dialysate pump 0ml/kg/min, waste pump 20ml/kg/min, plasma exchange 1 hour) plus plasma-filtration adsorption(PFA) (Blood pump: 120ml/min, Plasma separation rate 25-30%, PFA with acute multitherapeutic system (AMPLYA™ Italy) ≥30ml/min) and High volume plasma diafiltration (HVPDF) with CUREFLO™(ACF180W Japan) or Ultraflux® (AV1000S Fresenius Germany) , Blood pump same as PFA , replacement fluid pump 2000ml/h, dialysate pump 2000ml/h, waste pump 4000ml/h),with PFA and HVPDF for 15 hours in the first 3 days. If hemodynamically unstable or acute kidney injury(AKI) stage 2or 3,continue High volume hemofiltration(HVHF).Same protocol with control group after 3days.
  Interventions: Procedure: PEAF
- Control group (No Intervention): HVHF for septic shock with MODS is permitted in Control group routinely（Blood pump: 200ml/min, replacement fluid pump 45ml/kg/min, dialysate pump 45ml/kg/min, waste pump 90ml/kg/min, and high-volume hemofiltration for 16 hours with CUREFLO™(ACF180W Japan) or Ultraflux® (AV1000S Fresenius Germany) in the first 3 days after randomization.If hemodynamically unstable or AKI stage 2or 3,continue HVHF.

INTERVENTIONS:
Procedure: PEAF — PEAF that is therapeutic plasma exchange (TPE) with 20ml/kg/d Fresh frozen plasma (Blood pump: 120ml/min, replacement pump 20ml/kg/min, dialysate pump 0ml/kg/min, waste pump 20ml/kg/min, plasma exchange 1 hour) plus plasma filtration adsorption (PFA ) with acute multitherapeutic system( AMPLYA™ ITALY) ≥30ml/min lasting 15 hours plus High volume plasma diafiltration (HVPDF) with CUREFLO™(ACF180W Japan) or Ultraflux® (AV1000S Fresenius Germany) Blood pump: 120ml/min, replacement fluid pump 2000ml/h, dialysate pump 2000ml/h, waste pump 4000ml/h,and with high-volume plasma diafiltration for 15 hours）in the first 3 days. the treatment after three days later is same as the control group.
  Arms: PEAF

SUMMARY:
The purpose of this study is to evaluate the efficacy of coupled therapeutic plasma exchange adsorption diafiltration (PEAF )for treating septic shock with multiple organ dysfunction syndrome patients in ICU.

DETAILED DESCRIPTION:
Septic shock with multiple organ dysfunction syndrome (MODS) is a life-threatening clinical condition due to coagulant disorder immunoparalysis to infection. For this reason the extracorporeal therapies for the treatment of septic shock with MODS have become widespread in the ICU and, at the same time, new extracorporeal depurative techniques have been developed for the removal of inflammatory mediators. One of these techniques is therapeutic plasma exchange (TPE) that remove pathologically elevated cytokines and simultaneously to replace protective plasmatic factors. other techniques is coupled plasma-filtration adsorption (CPFA) that uses a sorbent once the separation between plasma and blood has been obtained with a plasma filter. The others is Plasma dialysis filtration(PDF) that can remove inflammatory mediators for patients with multiple organ dysfunction syndrome.The purpose of this study is to evaluate the efficacy of PEAF (coupled therapeutic plasma exchange adsorption diafiltration )for treating septic shock with multiple organ dysfunction syndrome patients in ICU.

ELIGIBILITY:
Inclusion Criteria:

1. Age, gender: 18-75 years old, male or female;
2. basic conditions: 20 ≤ APACHE II score ≤ 35 points and 10 ≤ Sequential Organ Failure Assessment(SOFA)≤ 18 points;
3. septic shock : On the basis of sepsis, after adequate fluid resuscitation, sustained hypotension requires maintenance of vasoactive drugs, mean arterial pressure（MAP）≥ 60 mmHg and Lactate ≥ 2.0 mmol/L; MODS: if the patient's SOFA score is ≥2 points, it means there is organ dysfunction. When the patient has two or more organ dysfunctions, it is MODS.

Exclusion Criteria:

1. can not remove the cause (surgical patients refused surgery, pan drug resistant infection without drug use)
2. Allergic to AMPLYA™ series
3. Presence of relative or absolute contraindications to PFA
4. MODS caused by severe liver disease
5. malignant tumors
6. Chronic end-stage disease (predicted to survive no more than one month)
7. Maternal and possibly pregnant women
8. participated in drug clinical trials within three months
9. Admission from an other ICU where the patient remained for more than 24 hours

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality within 28 days after randomization | 28 days after randomization
  efficacy

SECONDARY OUTCOMES:
All-cause mortality within 90 days from randomization | 90 days from randomization
  efficacy
free hours of vasoactive drugs from randomization | 14 days after randomization
  efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Ming Wu, MD, Principal Investigator — Shenzhen Second People's Hospita
Locations (12):
- China (12):
  - Dongguan Fifth People's Hospital (Taiping Hospital), Dongguan, Guangdong
  - Guangzhou General Hospital of Guangzhou Military Region, Guangzhou, Guangdong
  - School of Public Health, Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Luohu People's hospitial, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The eighth affiliated hospital, Sun Yat-Sen university, Shenzhen, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen Sixth People's Hospital (Nanshan Hospital), Shenzhen, Guangdong
  - Affiliated Baoan Hospital of Shenzhen, Southern Medical University (People' hospital of Baoan District), Shenzhen, Guangdong
  - Shenzhen Longgang Central Hospital, Shenzhen, Guangdong
  - Shenzhen hospital of southern medicial university, Shenzhen, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen

REFERENCES:
- [Background] Schwartz J, Padmanabhan A, Aqui N, Balogun RA, Connelly-Smith L, Delaney M, Dunbar NM, Witt V, Wu Y, Shaz BH. Guidelines on the Use of Therapeutic Apheresis in Clinical Practice-Evidence-Based Approach from the Writing Committee of the American Society for Apheresis: The Seventh Special Issue. J Clin Apher. 2016 Jun;31(3):149-62. doi: 10.1002/jca.21470. PMID 27322218
- [Result] Livigni S, Bertolini G, Rossi C, Ferrari F, Giardino M, Pozzato M, Remuzzi G; GiViTI: Gruppo Italiano per la Valutazione degli Interventi in Terapia Intensiva (Italian Group for the Evaluation of Interventions in Intensive Care Medicine) is an independent collaboration network of Italian Intensive Care units. Efficacy of coupled plasma filtration adsorption (CPFA) in patients with septic shock: a multicenter randomised controlled clinical trial. BMJ Open. 2014 Jan 8;4(1):e003536. doi: 10.1136/bmjopen-2013-003536. PMID 24401721
- [Result] Colomina-Climent F, Gimenez-Esparza C, Portillo-Requena C, Allegue-Gallego JM, Galindo-Martinez M, Molla-Jimenez C, Anton-Pascual JL, Rodriguez-Serra M, Martin-Ruiz JL, Fernandez-Arroyo PJ, Blasco-Ciscar EM, Canovas-Robles J, Herrera-Murillo M, Gonzalez-Hernandez E, Sanchez-Moran F, Solera-Suarez M, Torres-Tortajada J, Nunez-Martinez JM, Martin-Langerwerf D, Herrero-Gutierrez E, Sebastian-Munoz I, Palazon-Bru A, Gil-Guillen VF. Mortality Reduction in Septic Shock by Plasma Adsorption (ROMPA): a protocol for a randomised clinical trial. BMJ Open. 2016 Jul 12;6(7):e011856. doi: 10.1136/bmjopen-2016-011856. PMID 27406647
- [Result] Franchi M, Giacalone M, Traupe I, Rago R, Baldi G, Giunta F, Forfori F. Coupled plasma filtration adsorption improves hemodynamics in septic shock. J Crit Care. 2016 Jun;33:100-5. doi: 10.1016/j.jcrc.2016.02.005. Epub 2016 Feb 15. PMID 26975736
- [Result] Hazzard I, Jones S, Quinn T. Coupled plasma haemofiltration filtration in severe sepsis: systematic review and meta-analysis. J R Army Med Corps. 2015 Dec;161 Suppl 1:i17-i22. doi: 10.1136/jramc-2015-000552. PMID 26621809
- [Result] Yaroustovsky M, Abramyan M, Krotenko N, Popov D, Plyushch M, Rogalskaya E. A pilot study of selective lipopolysaccharide adsorption and coupled plasma filtration and adsorption in adult patients with severe sepsis. Blood Purif. 2015;39(1-3):210-217. doi: 10.1159/000371754. PMID 25765778
- [Result] Zhou N, Li J, Zhang Y, Lu J, Chen E, Du W, Wang J, Pan X, Zhu D, Yang Y, Chen Y, Cao H, Li L. Efficacy of coupled low-volume plasma exchange with plasma filtration adsorption in treating pigs with acute liver failure: A randomised study. J Hepatol. 2015 Aug;63(2):378-87. doi: 10.1016/j.jhep.2015.03.018. Epub 2015 Mar 24. PMID 25814048
- [Result] Berlot G, Agbedjro A, Tomasini A, Bianco F, Gerini U, Viviani M, Giudici F. Effects of the volume of processed plasma on the outcome, arterial pressure and blood procalcitonin levels in patients with severe sepsis and septic shock treated with coupled plasma filtration and adsorption. Blood Purif. 2014;37(2):146-51. doi: 10.1159/000360268. Epub 2014 Apr 26. PMID 24777037

DOCUMENTS (2):
  • Study Protocol (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT03589378/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT03589378/SAP_001.pdf